CLINICAL TRIAL: NCT02677337
Title: Novel Educational Interventions for Community Oncologists & Patients: Optimizing Renal Cell Carcinoma Outcomes Through Engagement
Brief Title: NCCN Renal Cell Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00065849
Record Dates: First submitted 2016-02-03; First posted 2016-02-09 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention)
- Educational Program (Other): chart abstraction will be conducted post education intervention component.
  Interventions: Other: chart abstraction; Other: Educational Program

INTERVENTIONS:
Other: chart abstraction — chart abstraction will be conducted pre and post education intervention to assess efficacy of education at point of care
  Arms: Educational Program
Other: Educational Program
  Arms: Educational Program

SUMMARY:
This study will consist of three parts: 1) a retrospective chart review of patients treated for mRCC from July 2013 until the start of the educational intervention; 2) an educational program for DCN community oncology providers and DCN community patients with mRCC, lasting 8 - 10 months, and 3) a second retrospective chart review of patients treated for mRCC starting at the time of the educational intervention until the intervention is completed.

DETAILED DESCRIPTION:
The initial retrospective cohort will serve as the pre-education control, and the second cohort will be the experimental group to assess the efficacy of the educational intervention to change care of patients with mRCC.

Chart Reviews. This study will begin with a multi-site chart review conducted at the Duke Cancer Network affiliated sites. The chart review will begin in late fall, 2015. The Duke Cancer Network team will perform chart abstraction for this study, with a goal of reviewing at least 60 charts of patients treated between July 2013 and October 2015.

The second data collection period will collect data on patients with mRCC seen at DCN sites after the date in fall 2015 when the educational intervention is rolled out. The target will again be at least 60 charts of patients treated during the time the educational intervention is actively available.

ELIGIBILITY:
Inclusion Criteria:

* Oncology providers (physicians, nurse practitioners, physicians' assistants) at DCN affiliated sites will be invited to use the performance support system and participate in the online virtual tumor boards for CME credit.

Exclusion Criteria:

* Non DCN affiliated sites providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assignment of patient to appropriate firstline treatment based on Heng Risk criterion | eight to ten months
  Improvement in the percentage of patients receiving appropriately prescribed first line therapy for metastatic renal cell cancer (mRCC)

SECONDARY OUTCOMES:
Percentage of increase in duration of treatment with appropriate first line therapy | eight to ten months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Criscione-Schreiber, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
This trial may potentially be published.